CLINICAL TRIAL: NCT06208085
Title: An Avocado Intervention to Increase the Nutrients in Human Milk in Support of Infant Cognitive Development
Brief Title: Avocado Consumption, Nutrients in Human Milk, and Infant Cognitive Development
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Avocado Nutrition Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-2933
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Breastfeeding, Exclusive
Keywords: Breastfeeding; Avocados; Infant cognition
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to avocado or no avocado groups. The avocado group will be asked to consume an avocado a day for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avocado (Experimental): Participants will be provided avocados and asked to consume an avocado a day for 12 weeks.
  Interventions: Dietary Supplement: Avocado
- No Avocado (No Intervention): Comparison arm in which no intervention occurs.

INTERVENTIONS:
Dietary Supplement: Avocado — Intervention arm
  Arms: Avocado

SUMMARY:
The goal of this interventional study is to establish a whole food, avocado, as a viable study material to supplement mothers and infants with nutrients that support optimal brain development. Eighty-eight breastfeeding dyads, 3m postnatal, will participate in this study designed to:

1. To document whether lactating mothers will comply in the consumption of 5 avocados a week for 12 weeks.
2. To ascertain the choline, lutein, and fatty acids present in human milk in women who eat avocado.
3. To measure the cognitive advantage conferred to infants whose mothers consume avocados while breastfeeding compared to a non-avocado-eating reference group.

To this end, healthy, lactating women who are 13 weeks postpartum and their infants will be enrolled. Mothers will be provided avocados on a bi-weekly basis and will be asked to consume an avocado a day. Infant cognition will be tested when the infants are 4.5 and 6 months of age. Milk samples and diet data will be collected and assayed on a bi-weekly basis.

DETAILED DESCRIPTION:
Nutrients do not appear in nature alone with some appearing together more often than not. It is reasonable to posit that nutrients are working together, and thus, the synergies among the nutrients are important to understand. First, choline is integral to brain fatty acids in that phosphatidylcholine (PC) serves an active role in mediating hepatic export of fatty acids to extra-hepatic tissues such as brain: fatty acids are stored in the liver, and PC moves them to the brain. Erythrocyte PC-DHA is integral to our consideration of a potential mechanism behind our results. Enriched in docosahexaenoic acid (DHA), PC comprises the cell membrane and influences membrane fluidity with downstream effects on signal transduction thereby improving speed of processing and recognition memory. Lutein has a very important role also in that it is known to co-localize with DHA specifically resulting in improvements in visual acuity, for example, and in general, it has been shown to protect fatty acids from peroxidation. Indeed, interventions with avocado have shown a significant increase in plasma lutein and a decrease in lipid peroxidation. It is hypothesized that lutein is also having this effect in the brain. As work with single nutrient supplementation does not yield strong cognitive effects, the investigators study the effects of co-occurring nutrients on cognitive development. The proposed study is designed to achieve an overall objective of establishing a whole food, avocado, as a viable study material in the pursuit of optimization of human milk with nutrients that support brain development. The long-term goal is to establish guidelines for maternal nutrition during gestation and lactation that include key nutrients for fetal and infant brain development, and the overall impact of this research program will be to set children on a trajectory for school readiness. The central hypothesis is that maternal avocado consumption will provide nutrients through human milk to support the development and function of neural substrates that support cognition. Specifically, choline, lutein, and fatty acids will work synergistically to improve brain function.

Mothers will be randomized to avocado or no avocado (due to lack of an appropriate control food). Participants will come to the lab 3 times across 6 months (enrollment/3months, 4.5 months, and 6 months). Milk sample will be provided every two weeks and will be picked up from the participants. At pickup, the avocado group will also be provided a new supply of avocados. Diet data will be collected at each visit/pickup (every two weeks). The infant will complete a recognition memory test using electrophysiology at 6 months as well as the Bayley Scales of Infant Development at 4.5 months. The mother will complete a temperament questionnaire at 3 and 6 months. Saliva samples will also be collected.

ELIGIBILITY:
Inclusion Criteria

* Healthy lactating women at 13 weeks postpartum
* Planning to exclusively breastfeed to 6 months of age
* Gave birth at 38 weeks or greater gestation without remarkable incident
* Pre-pregnancy BMI <30

Exclusion Criteria

* Gestational diabetes
* Infant with diagnosis or documented suspicion of developmental delay
* Any documented seizure activity in infant
* Family history of avocado, latex, or banana allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recognition Memory in an Oddball Task | Week 12 (at 6 months of age)
  The difference in microvolts between the negative deflection to novel pictures and the negative deflection to familiar pictures at approximately 100-400ms after the pictures come on the screen will be measured in an event-related potentials (ERP) paradigm. The investigators hypothesize that the avocado group will have better memory for the familiar pictures than the no avocado group.
Change in Choline Content of Milk | Baseline, Week 12
  Human milk will be assayed for choline every two weeks and analyzed for change over time (7 data points across 12 weeks).
Change in Lutein Content of Milk | Baseline, Week 12
  Human milk will be assayed for lutein every two weeks and analyzed for change over time (7 data points across 12 weeks).
Change in Fatty Acid Content of Milk | Baseline, Week 12
  Human milk will be assayed for fatty acids every two weeks and analyzed for change over time (7 data points across 12 weeks).

SECONDARY OUTCOMES:
Bayley Scales of Infant Development (BSID) | Week 6 (at 4.5 months of age)
  Neurodevelopmental assessment scores are age dependent and based motor and behavioral abilities, often reported for normal or abnormal for age. Bayley Scales of Infant and Toddler Development, 3rd edition, (Bayley III) is an instrument designed to measure the developmental functioning of infants and toddlers between the ages of 1 month and 42 months (age adjustments for prematurity are accommodated with the tool). It provides age specific composite scores for cognitive (91 items, score min 55 max 145), language (98 items, score min 47 max 153), and motor (138 items, score min 46 max 154) skills. For all scales, higher scores are better and lower scores indicate possible delay/deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Nutrition Research Institute, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
To ensure long-term findability, accessibility, interoperability, and reusability, the de-identified data from participants who agree to sharing and the codebook will be deposited in the UNC Dataverse, a generalist data repository managed by the Odum Institute at the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be made available in University of North Carolina at Chapel Hill (UNC) Dataverse at the time of associated publication or end of the performance period, whichever comes first. Data will be stored and available in UNC Dataverse in perpetuity as indicated in UNC Dataverse preservation policies.
Access Criteria: Interested researchers who email their interest will be granted access on a case-by-case basis after agreement between the funder and the PI, who co-own the data.
URL: https://dataverse.unc.edu/